CLINICAL TRIAL: NCT04589780
Title: Is There a Relationship Between the Risk of Injury and Posture in Wrestlers?
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-38/364
Record Dates: First submitted 2020-10-10; First posted 2020-10-19 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Sport Injury; Posture; Wrestling; Risk Reduction
Keywords: Wrestling; Functional movement screen; Injury risk; Posture
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Posture Assessment: Posture will be assessed with New York Posture Rating Chart (NYPR) originally published in 1958
- Sagittal spinal alignment and mobility: Sagittal spinal alignment and mobility will be measured using the Spinal Mouse (IdiagAG Mülistrasse 18 CH-8320 Fehraltorf, Switzerland), a computer-aided, non-invasive device.
- Injury risk assessment: Injury risk will be evaluated with Functional Movement Screen (FMS) test battery. A previous systematic review has demonstrated acceptable reliability for the FMS

SUMMARY:
This study was planned to investigate the relationship between the risk of injury and posture in wrestlers. The study will be included male wrestlers. The spine posture and flexibility of the athletes will be measured during standing position with the Idiag M360® brand Spinal Mouse (SM), while the overall body posture will be measured from the anterior and lateral sides using the New York Posture Analysis Method (NYPAM). Injury risks of the athletes will be evaluated by Functional Movement Screen (FMS) which was consisting of seven basic movement patterns.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18 and 40
* To be a professional wrestler who won medals in the Turkey championships

Exclusion Criteria:

* had injury for in the last 6 months
* had a history of surgery, or chronic and progressive disease
* had any orthopaedic or neurological problems

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In this cross-sectional study, 18- to 40-year-old elite wrestler who have won medals in their championships from four different clubs will be tested
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Posture Assessment | 2 weeks
  Posture will be assessed with New York Posture Rating Chart (NYPR) originally published in 1958
Sagittal spinal alignment and mobility | 2 weeks
  Sagittal spinal alignment and mobility will be measured using the Spinal Mouse (IdiagAG Mülistrasse 18 CH-8320 Fehraltorf, Switzerland), a computer-aided, non-invasive device
Injury risk assessment | 2 weeks
  Injury risk will be evaluated with Functional Movement Screen (FMS) test battery. A previous systematic review has demonstrated acceptable reliability for the FMS

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No